CLINICAL TRIAL: NCT01878136
Title: Effect of Intraventricular tPA Following Aneurysmal Subarachnoid Hemorrhage
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Time constraints
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Stephan Munich, Neurosurgery Resident, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13011803
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm; Cerebral Aneurysm; Hydrocephalus
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Intracranial Aneurysm; Hydrocephalus | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraventricular tPA (Active Comparator): Tissue Plasminogen Activator (tPA)
  Dose: 1 mg Q8 hr x 12 doses, or until blood is cleared from the ventricles and cisterns Adminstration: Intraventricular; via previously placed external ventricular drain
  Interventions: Drug: Tissue Plasminogen Activator
- Placebo (Placebo Comparator): Placebo
  Dose 1 mL sterile saline
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — Dose: 1mg Q8 x 12 doses, or until clearance of blood from ventricles and cisterns Administration: intraventricular administration (through external ventricular drain)
  Other Names: Activase; Alteplase

SUMMARY:
This study will evaluate the hypothesis that the administration of intraventricular tPA reduces the rates of cerebral vasospasm and ventriculoperitoneal shunt-dependent hydrocephalus in patients with aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old.
* SAH due to aneurysm, as determined by CT angiogram or cerebral angiogram.
* Modified Fisher (mF) grade 3 or 4 SAH, defined as thick cisternal blood without (grade 3) or with (grade 4) intraventrciular blood.
* Exclusion of the aneurysm from the parent circulation by endovascular embolization (Raymond class I or II) within 48 hours of ictus.
* Ventriculostomy placement must occur prior to randomization.
* Informed consent obtained from the patient or patient's decision maker

Exclusion Criteria:

* Determination by treating physician(s) that no ventriculostomy is needed.
* Presence of intrinsic clotting disorders (e.g. due to hepatic failure, nephrotic syndrome, etc). Subjects whose pharmacologic anticoagulation is reversed, as determined by PT/INR, PTT within our institution's normal range, will be permitted to participate in this study.
* Presence of significant anemia, defined as hemoglobin < 8 gm/dL.
* Patients who undergo endovascular techniques requiring post-operative dual anti-platelet therapy.
* Residual aneurysm sac filling (Raymond class III occlusion).
* Aneurysm or vessel perforation during the endovascular procedure.
* Presence of craniectomy.
* Significant neurologic disability prior to the onset of SAH.
* Determination that administration of tPA/placebo cannot be initiated within 72 hours of symptom onset.
* Presence of untreated intracranial aneurysms larger than 3mm on CT angiography or cerebral angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Outcome | 1-60 days after SAH
  The composite primary outcome will consist of the rates of ventriculoperitoneal shunt (VPS) placement, clinically significant vasospasm, and death. VPS placement serves as surrogate measure of hydrocephalus. These outcomes will be measured during the patient's hospitalization.

SECONDARY OUTCOMES:
Rate of new intracranial hemorrhage | 1-14 days after SAH
  New intracranial hemorrhage will be defined as any new parenchymal or ventricular hemorrhage occurring after the first dose of study drug/placebo.
Rate of intracranial infection | 1-14 after SAH
  The presence of infection will require identification of an offending organism via CSF cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Munich, MD, Principal Investigator — Rush University Medical Center, Department of Neurosurgery; Roham Moftakhar, MD, Study Director — Rush University Medical Center, Department of Neurosurgery
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States